CLINICAL TRIAL: NCT01200888
Title: Differentiating Outcome Measures in Infants/Young Children With Cystic Fibrosis Utilizing Controlled Ventilation Infant/Young Child Chest CT Scanning and Lung Function Testing
Brief Title: Controlled Ventilation CT in CF Infants
Status: Terminated | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Terry Robinson, Associate Professor, Stanford University
Other Study IDs: SU-09092010-6830; eProt #17572
Record Dates: First submitted 2010-09-10; First posted 2010-09-14 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of the study is to implement a new method of performing chest CT imaging in young children with cystic fibrosis at Packard Children's Hospital. This technique will be used to evaluate early lung disease comparing quantitative chest CT air trapping and airway measurements with lung function measurements in infants, toddlers, and young children with chronic lung disease.

ELIGIBILITY:
Inclusion Criteria:

1. Infants and young children (age ~ 2/3 months to < 5 years)
2. Diagnosed with cystic fibrosis with either 2 identified CFTR gene mutations, or a positive sweat chloride
3. Informed consent by parent or legal guardian.
4. Ability to comply with study visit procedures as judged by the investigator.

Exclusion Criteria:

1. Acute wheezing and/or respiratory distress at either study visit.
2. Acute intercurrent respiratory infection, defined as an increase in cough, wheezing, or respiratory rate with onset in 1 week preceding Study visit.
3. Oxygen saturation < 90% on room air at study visit.
4. Any medical condition that in the opinion of the investigator precludes subject participation.

Ages: 2 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Young children with cystic fibrosis at Packard Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Quantitative Air Trapping, A2 & A3 | Baseline & F/U
  Quantitative Chest CT Air Trapping by CT post-processing for Measure A2 & Measure A3 (% of segmented total lung)
Quantitative CT Airway Measurements (AWT/TAD, LD/TAD, Wall Area %, Lumen Area % | Baseline & F/U
  Quantitative Chest CT airway measurements by CT Post-Processing. AWT/TAD = Airway Wall Thickness/Total Airway Diameter LD/TAD = Lumen Diameter/Total Airway Diameter Wall Area % = Wall Area/Total Airway Area (%)

SECONDARY OUTCOMES:
FEV 0.5 sec | Baseline & F/U
  FEV 0.5sec = % predicted
FEF 85% | Baseline & F/U
  FEF 85% (% predicted)
FEF25-75% | Baseline & F/U
  FEF25-75% (% predicted)

CONTACTS AND LOCATIONS:
Overall Officials: Terry Earl Robinson, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States